CLINICAL TRIAL: NCT05608278
Title: Four-day Intensive Treatment Versus Standard Cognitive Behavioral Therapy for Adults With Obsessive-compulsive Disorder: a Single-blind, Randomized Controlled Non-inferiority Trial
Brief Title: Four-day Intensive Treatment Versus Standard Cognitive Behavioral Therapy for Adults With Obsessive-compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Helse-Bergen HF (Other)
Responsible Party: Principal Investigator, Christian Rück, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCD - B4DT vs standard CBT
Record Dates: First submitted 2022-10-26; First posted 2022-11-08 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Cognitive Behavioral Therapy; Obsessive-Compulsive Disorder; Randomized Controlled Trial
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bergen 4-Day Treatment (B4DT) (Experimental): Patients in this arm will receive an intensive treatment delivered mostly in group format. The group sizes will be 3-6 participants with a 1:1 patient to therapist ratio. In the week before the intensive part of the treatment, participants will have two scheduled phone/video calls with a therapist. Day 1 (half-day) of the intensive treatment includes psychoeducation and deciding on exposure tasks. Days 2 and 3 (whole days) focus on individually tailored and therapist-assisted ERP in as many most relevant settings as possible. In the evenings, patients are encouraged to continue with self-guided ERP and may receive therapist support via text messages or phone calls on demand. On day 3, patients can invite relatives to a psychoeducation session. Day 4 (half-day) of the intensive treatment focuses on treatment summary and relapse prevention, as well as planning self-guided ERP for the upcoming 3 weeks.
  After 16 weeks, participants have individual follow-up sessions without ERP.
  Interventions: Behavioral: Bergen 4-Day Treatment (B4DT)
- Gold standard cognitive behavioral therapy (gold standard CBT) (Active Comparator): Patients will receive 16 sessions of individual CBT for OCD with an emphasis on ERP, delivered over a time period of 14 weeks according to a validated protocol. Sessions will be held twice weekly at a specialist clinic during the first 2 weeks and once a week for the remaining 12 weeks. Sessions 1-2 contain psychoeducation about OCD and CBT, goal setting, and planning of ERP exercises. Sessions 3-14 include therapist-guided ERP (at the clinic, in the patients' homes or elsewhere as needed) with planned self-practice ERP between sessions. Sessions 15-16 contain a summary of the treatment and lessons learned, as well as relapse prevention and planning of continued self-practice ERP.
  Interventions: Behavioral: Gold standard cognitive behavioral therapy (gold standard CBT)

INTERVENTIONS:
Behavioral: Bergen 4-Day Treatment (B4DT) — Novel CBT treatment
  Arms: Bergen 4-Day Treatment (B4DT)
Behavioral: Gold standard cognitive behavioral therapy (gold standard CBT) — Gold standard CBT treatment
  Arms: Gold standard cognitive behavioral therapy (gold standard CBT)

SUMMARY:
The goal of this clinical trial is to compare a novel, condensed version of cognitive behavioral therapy (Bergen 4-Day Treatment, B4DT) to the gold standard psychological treatment (gold-standard CBT) for obsessive compulsive disorder (OCD).

The main question it aims to answer is:

• Is B4DT non-inferior to standard cognitive behavioral therapy (CBT) with regard to OCD symptoms 14 weeks after treatment start?

Adult patients with obsessive compulsive disorder will be randomly assigned to receive either gold standard CBT one to two times per week for 14 weeks, or 4 days of B4DT during one week.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder is a persistent and disabling psychiatric disorder. Individual cognitive behavioral therapy (CBT) with exposure and response prevention (ERP) is an effective treatment for OCD and is recommended as a first-line intervention. However, patients need to remain in treatment for several months and even after that, around 50% remain symptomatic despite this lengthy treatment. In response to this, a novel, condensed version of CBT, B4DT, has been developed. B4DT has shown promising results in several uncontrolled trials and one randomized controlled trial with inactive control, however it has yet to be directly compared to gold-standard individual CBT.

This single blind, randomized controlled trial with 120 patients (60 per arm) will compare B4DT to gold standard CBT. The primary outcome is the blind-rater administered Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). The investigators hypothesize that B4DT will be non-inferior to gold standard CBT 14 weeks after treatment start. The non-inferiority margin is set at 4 points on the Y-BOCS.

Secondary outcomes are cost effectiveness, speed of response, response and remission rates, dropout rate, and negative effects. The investigators hypothesise that participants that receive B4DT will improve faster than patients that receive standard CTB, but for the rest of the secondary outcomes, the investigators have no directed hypotheses.

A more detailed preregistration, and all analysis scripts, are available at Open Science Framework (https://osf.io/w5bfp/).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Primary diagnosis of OCD according to the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5).
3. Clinician-rated Y-BOCS score of ≥ 16
4. Written informed consent.
5. To be willing and able to attend treatment at any one of the two treatment clinics, regardless of the clinic where the initial assessment took place (the two clinics are located at different locations in Stockholm, about 20 Km apart).
6. Be fluent in Swedish.

Exclusion Criteria:

1. Other psychological treatment for OCD planned during trial period.
2. Completed CBT with ERP for OCD in the last 12 months.
3. Changes in psychotropic medication within the last 2 months.
4. Bipolar disorder.
5. Psychosis.
6. Alcohol or substance dependence.
7. Organic brain disorder.
8. Hoarding disorder or OCD with primary hoarding symptoms.
9. Suicidal ideation that would warrant close monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (Y-BOCS), clinician-administered | Change from baseline to 14 weeks after treatment start. Additional measures at week 4 and 7, and at the 7- and 16-month follow-up
  Clinician administered scale that measures the severity of obsessions and compulsions. Ten questions, with scores ranging from 0 to 4 (most severe), address time, interference, distress, resistance and control over obsessions and compulsions (total score range from 0 to 40).

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S) | 14 weeks after treatment start. Additional measures at week 4 and 7, and at the 7- and 16-month follow-up
  Used to assess rates of response and remission. The Clinical Global Impression - Severity (CGI-S) and Clinical Global Impression - Improvement (CGI-I) Scales will be used to assess overall clinical severity and consequent treatment response (scores of "very much improved" (1) or "much improved" (2) will define treatment response according to previous trials in tic disorders.
Clinical Global Impression - Improvement (CGI-I) | 14 weeks after treatment start. Additional measures at week 4 and 7, and at the 7- and 16-month follow-up
  Used to assess rates of response and remission. The Clinical Global Impression - Severity (CGI-S) and Clinical Global Impression - Improvement (CGI-I) Scales will be used to assess overall clinical severity and consequent treatment response (scores of "very much improved" (1) or "much improved" (2) will define treatment response according to previous trials in tic disorders.
Dropout rate in both arms | Gold standard CBT: week 15. B4DT: week 3.
  A dropout will be defined as a patient in the B4DT arm that participates in less than 1.5 full days at the clinic, or a patient in the gold standard CBT arm that participates in less than 8 CBT sessions.
Treatment Inventory of Costs in Psychiatric Patients (TIC-P) | Pre-treatment, at week 15, and at the 7- and 16-month follow-ups
  Self-rated questionnaire on healthcare utilization and productivity losses in patients with a psychiatric disorder. The TIC-P questionnaire measures costs in two dimensions: use of health resources and loss of productivity. Lower cost is better.
Negative Effects Questionnaire (NEQ) | 14 weeks after treatment start. Additional measures at the 7- and 16-month follow-ups
  Self-rated questionnaire on negative effects. It contains 32 items that are scored on a five point Likert-scale (0-4) and differentiates between negative effects that are attributed to treatment and those possibly caused by other circumstances. The total score of the NEQ ranges from 0 to 80 points, a higher score reflects more negative effects.
Assessing Quality of Life 6 Dimensions (AQoL-6D) | Change from baseline to 14 weeks after treatment start. Additional measures at the 7- and 16-month follow-ups
  Used to assess cost-effectiveness. 20 questions that assess different aspects of quality of life. The AQoL provides a utility score that ranges from 1.00 (full health) to 0.00 (death-equivalent health states) to -0.04 (health states worse than death).

OTHER OUTCOMES:
Patient Exposure/Response Prevention Adherence Scale (PEAS) | Gold standard CBT: week 4, 7, and 15. B4DT: week 3.
  Measures the patient's between-session adherence to the therapist's exposure and response prevention instructions. The scale has three subscales: exposure assignments attempted, the quality of exposure assignments attempted, and the percentage of rituals resisted between session. Each subscale ranges from 0 to 100%, high scores represent better adherence.
Yale-Brown Obsessive Compulsive Scale-Self-Rated (Y-BOCS-SR) | Pre-treatment, at week 15, and at the 7- and 16-month follow-ups
  Self rated version of the primary outcome that measures severity of obsessions and compulsions. It consists of 10 items rated on a 5-point Likert scale (0 to 4) with higher scores denoting greater symptom severity.
Montgomery-Åsberg Depression Rating Scale-Self-Rated (MADRS-S) | Pre-treatment, at week 15, and at the 7- and 16-month follow-ups
  Measures symptom severity of depression. MADRS is a 9-item depressive symptoms scale where the symptoms are assessed on a 7-point likert scale from no symtoms to very high severity. The total score ranges from 0 to 54 with higher score indicating more severe problems.
Work and Social Adjustment Scale (WSAS) | Pre-treatment, at week 15, and at the 7- and 16-month follow-ups
  Measures impairment in functioning. Scores range from 0-40, with lower scores representing better functioning.
Credibility/Expectancy Questionnaire (CEQ) | Week 2
  Measures treatment expectancy and rationale credibility. The CEQ is a 5-item measure of the treatment's credibility and the patients' expectations. The patients assess each domain on a 11-point likert scale (scored 0-10), with a total score ranging between 0-50 where higher score indicates higher credibility and higher expectations.
Working Alliance Inventory-Short Form Revised (WAI-SR) | Week 2
  Measures the therapeutic alliance in therapy. The WAI-SR is a 12-item measure of the patient's experience of their working alliance with the therapist. The patients assess each item on a 7-point likert scale (scored 0-6), with a total score ranging between 0-72 where higher score indicates higher better working alliance according to the patient.
Obsessive-Compulsive Inventory-Revised (OCI-R) | Pre-treatment, at week 15, and at the 7- and 16-month follow-ups
  Self-rating scale that measures the severity and type of symptoms of OCD. The Obsessive-Compulsive Inventory-Revised (OCI-R) has 18 items. Each item is scored on a 5 point scale from 0 to 4. Total score ranges from 0 to 72, higher scores represent more severe OCD.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Psykiatri Nordväst, Stockholms Läns Sjukvårdsområde (SLSO), Stockholms Läns Landsting, Stockholm
  - Psykiatri sydväst, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be shared through a searchable database, Swedish national data service (SND), with restricted access. Only meta-data will be shared without restrictions. Researchers that want access to the raw data data will have to submit an additional application an ethical review board.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The supporting information will become available for everybody on Open Science Framework (https://osf.io/w5bfp/) before inclusion of the first participant. We will not delete anything, potential changes will be transparently reported through time stamped documents.
  We plan to submit the raw data to SND after completion. We will never delete it.
Access Criteria: Approved ethics application.
URL: https://snd.gu.se/en

REFERENCES:
- [Derived] Ivanova E, Fondberg R, Flygare O, Sannemalm M, Asplund S, Dahlen S, Sampaio F, Andersson E, Mataix-Cols D, Ivanov VZ, Ruck C. Study protocol for a single-blind, parallel-group, randomised, controlled non-inferiority trial of 4-day intensive versus standard cognitive behavioural therapy for adults with obsessive-compulsive disorder. BMJ Open. 2023 Dec 14;13(12):e076361. doi: 10.1136/bmjopen-2023-076361. PMID 38101824

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT05608278/Prot_SAP_000.pdf